CLINICAL TRIAL: NCT06169371
Title: Abemaciclib Dose Escalation to Maintain Intensity (ADE-MI)
Acronym: BRE-09
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Vijayakrishna Krishnamurthy Gadi, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0433
Record Dates: First submitted 2023-11-28; First posted 2023-12-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm adjuvant abemaciclib (Other): Participants will receive adjuvant abemaciclib which will be dose escalated. Abemaciclib will be taken at 50 mg by mouth twice a day during Week 1, 100 mg by mouth twice a day during Week 2, and 150 mg by mouth twice a day starting Week 3.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Week 1 50mg orally BID
Drug: Abemaciclib — Week 2 100mg orally BID
Drug: Abemaciclib — Week 3+ 150mg orally BID

SUMMARY:
This is a post-marketing single arm, phase IV trial in which patients with high-risk early-stage HR+HER2- breast cancer will receive adjuvant abemaciclib in combination with endocrine therapy (ET) After study intervention, participants will remain on combination abemaciclib + ET at the discretion of their treating providers

DETAILED DESCRIPTION:
Dose escalation (DE) was shown to minimize the rates of Grade 3 diarrhea in the setting for HER2+ breast cancer. DE can improve tolerability for drugs such as abemaciclib. This is a post-marketing single arm, phase IV trial in which patients with high-risk early-stage HR+HER2- breast cancer will receive adjuvant abemaciclib in combination with endocrine therapy (ET) After study intervention, participants will remain on combination abemaciclib + ET at the discretion of their treating providers

In this study, the investigators we will test the hypothesis that gradual up-titration of abemaciclib dose over a course of 2-3 weeks will decrease the rate of G3 or worse diarrhea, permitting more patients to remain at the intended dose when evaluated at day 84

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2
* Histologically confirmed early-stage HR+HER2- breast cancer documented by biopsy who are prescribed adjuvant abemaciclib
* Able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
* Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Chronic history of diarrhea
* Active infection requiring systemic therapy
* Uncontrolled HIV/AIDS or active viral hepatitis
* Pregnant or nursing
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Other major comorbidity as determined by study PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Increase the proportion of subjects on FDA approved dose of Abemaciclib (150mg BID) at day 84 | Day 84
  Number of subjects that continue to receive Abemaciclib 150mg BID for 84 days

SECONDARY OUTCOMES:
How many days with Grade 2 or greater of diarrhea in the first month | 1 month
  Number of days with Grade 2 or greater in the first month
Rate of Grade 3 or greater of diarrhea in the first 3 months | 3 months
  Nuber of subjects who experienced Grade 3 or greater by the total number of subjects enrolled
Disease Free Survival (DFS) | 1 year
  Number of subjects that have DFS from D1 of treatment until the criteria for disease progression as defined by RECIST 1.1 or death
Disease Free Survival (DFS) | 2 years
  Number of subjects that have DFS from D1 of treatment until the criteria for disease progression as defined by RECIST 1.1 or death
Overall Survival (OS) | 1 year
  OS is defined as the time from D1 of treatment until death
Overall Survival (OS) | 2 years
  OS is defined as the time from D1 of treatment until death
Overall Survival (OS) | 3 years
  OS is defined as the time from D1 of treatment until death
Subject reported outcomes regarding adverse events | 5 years
  Toxicity grade as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: VK Gadi, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois, Chicago, Illinois
  - Iowa Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No